CLINICAL TRIAL: NCT06520904
Title: Effect of PCSK9 Inhibitors on Coronary Atherosclerotic Plaques Derived From Optical Coherence Tomography in Patients With Premature Coronary Artery Disease: a Randomized Controlled Trial
Brief Title: Effect of PCSK9 Inhibitors on Coronary Atherosclerotic Plaques Derived From Optical Coherence Tomography
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Zhenyan Fu, PHD, Principle Investigator, First Affiliated Hospital of Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPCAP-OCT
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Optical Coherence Tomography
Keywords: Coronary Artery Disease; Lipid-lowering Therapy; PCSK9; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9 inhibitor group (Experimental): PCSK9 Inhibitors Combined with Moderate-Intensity Statin Therapy
  Interventions: Drug: PCSK9 inhibitor
- Intensive statin group (Other): Intensive statin therapy
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: PCSK9 inhibitor — PCSK9 inhibitors combined with moderate-intensity statin therapy
  Arms: PCSK9 inhibitor group
Drug: Statin — Intensive statin therapy
  Arms: Intensive statin group

SUMMARY:
The presence of coronary atherosclerotic vulnerable plaque significantly impacts the clinical outcomes of patients diagnosed with coronary artery disease (CAD). However, the influence of PCSK9 inhibitors on stabilizing coronary atherosclerotic plaques in individuals with early-onset CAD, evaluated through optical coherence tomography (OCT), remains inadequately understood. Moreover, there is a notable absence of relevant randomized controlled trials investigating this phenomenon. This current study represents a single-center, randomized, controlled, open-label trial conducted among Asian patients with early-onset CAD. Its principal objective was to explore the effects of PCSK9 inhibitors on coronary atherosclerotic plaque morphology as assessed by OCT.

DETAILED DESCRIPTION:
Following initial percutaneous coronary intervention (PCI) for culprit lesions in patients with early-onset coronary artery disease (CAD) and ≥2 additional lesions meeting baseline lipid criteria, optical coherence tomography (OCT) was employed to evaluate non-culprit lesion sites for detailed characterization of plaque features including calcification, fibrosis, fibrolipid deposition, necrosis, minimum fibrous cap thickness (mFCT), and maximum lipid arc (MLA). Subsequently, patients were randomized in a 1:1 ratio to receive either intensive statin therapy alone or a combination of PCSK9 inhibitor with moderate-intensity statin therapy, using a random number allocation method. After 1 year of treatment and follow-up, OCT reassessment of non-culprit vessel critical lesions was conducted, documenting plaque characteristics such as calcification, fibrosis, fibrolipid content, necrosis, as well as stability parameters like mFCT and MLA at lesion sites. OCT findings were compared longitudinally within each treatment group and between groups receiving PCSK9 inhibitor combined with statin therapy versus intensive statin therapy alone. Baseline clinical profiles, biochemical markers, imaging findings, and incidence of adverse cardiovascular events during the follow-up period were also meticulously recorded for all enrolled early-onset CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-55 years and women aged 18-65 years;
* CAD patients with coronary angiographically confirmed lesions in ≥2 vessels; at least one vessel was critically diseased (50-70% stenosis level);
* LDL-C >3.4 mmol/L without regular statin therapy or LDL-C >1.8 mmol/L after 4 weeks of statin lipid-lowering therapy.

Exclusion Criteria:

* Known allergies or contraindications to PCSK9 inhibitors and/or statin therapy;
* Prior use of PCSK9 inhibitors;
* Prior history of hemorrhagic stroke;
* Prior coronary artery bypass grafting or coronary intervention;
* Inability to perform OCT imaging or unclear imaging;
* Severe renal insufficiency (creatinine clearance < 30 mL/min);
* Severe hepatic dysfunction;
* Baseline triglycerides > 5.6 mmol/L;
* Pregnant or lactating women;
* Life expectancy not exceeding 1 year;
* In the judgment of the investigator, unsuitable for this study for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mFCT | Immediate and 1 year after PCI
  minimum fibrous cap thickness
MLA | Immediate and 1 year after PCI
  maximum lipid arc
Calcification | Immediate and 1 year after PCI
  calcification
Fibrosis | Immediate and 1 year after PCI
  fibrosis
Fibrolipid deposition | Immediate and 1 year after PCI
  fibrolipid deposition
Necrosis | Immediate and 1 year after PCI
  necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyan Fu, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No
IPD will be made available on reasonable request to the official agencies.

REFERENCES:
- [Background] Johnson TW, Raber L, di Mario C, Bourantas C, Jia H, Mattesini A, Gonzalo N, de la Torre Hernandez JM, Prati F, Koskinas K, Joner M, Radu MD, Erlinge D, Regar E, Kunadian V, Maehara A, Byrne RA, Capodanno D, Akasaka T, Wijns W, Mintz GS, Guagliumi G. Clinical use of intracoronary imaging. Part 2: acute coronary syndromes, ambiguous coronary angiography findings, and guiding interventional decision-making: an expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. Eur Heart J. 2019 Aug 14;40(31):2566-2584. doi: 10.1093/eurheartj/ehz332. PMID 31112213
- [Background] Mortensen MB, Dzaye O, Steffensen FH, Botker HE, Jensen JM, Ronnow Sand NP, Kragholm KH, Sorensen HT, Leipsic J, Maeng M, Blaha MJ, Norgaard BL. Impact of Plaque Burden Versus Stenosis on Ischemic Events in Patients With Coronary Atherosclerosis. J Am Coll Cardiol. 2020 Dec 15;76(24):2803-2813. doi: 10.1016/j.jacc.2020.10.021. PMID 33303068
- [Background] Taron J, Foldyna B, Mayrhofer T, Osborne MT, Meyersohn N, Bittner DO, Puchner SB, Emami H, Lu MT, Ferencik M, Pagidipati NJ, Douglas PS, Hoffmann U. Risk Stratification With the Use of Coronary Computed Tomographic Angiography in Patients With Nonobstructive Coronary Artery Disease. JACC Cardiovasc Imaging. 2021 Nov;14(11):2186-2195. doi: 10.1016/j.jcmg.2021.03.019. Epub 2021 Apr 14. PMID 33865792
- [Background] Koskinas KC, Ughi GJ, Windecker S, Tearney GJ, Raber L. Intracoronary imaging of coronary atherosclerosis: validation for diagnosis, prognosis and treatment. Eur Heart J. 2016 Feb 7;37(6):524-35a-c. doi: 10.1093/eurheartj/ehv642. Epub 2015 Dec 11. PMID 26655874
- [Background] Prati F, Romagnoli E, Gatto L, La Manna A, Burzotta F, Ozaki Y, Marco V, Boi A, Fineschi M, Fabbiocchi F, Taglieri N, Niccoli G, Trani C, Versaci F, Calligaris G, Ruscica G, Di Giorgio A, Vergallo R, Albertucci M, Biondi-Zoccai G, Tamburino C, Crea F, Alfonso F, Arbustini E. Relationship between coronary plaque morphology of the left anterior descending artery and 12 months clinical outcome: the CLIMA study. Eur Heart J. 2020 Jan 14;41(3):383-391. doi: 10.1093/eurheartj/ehz520. PMID 31504405
- [Background] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Background] Raber L, Koskinas KC, Yamaji K, Taniwaki M, Roffi M, Holmvang L, Garcia Garcia HM, Zanchin T, Maldonado R, Moschovitis A, Pedrazzini G, Zaugg S, Dijkstra J, Matter CM, Serruys PW, Luscher TF, Kelbaek H, Karagiannis A, Radu MD, Windecker S. Changes in Coronary Plaque Composition in Patients With Acute Myocardial Infarction Treated With High-Intensity Statin Therapy (IBIS-4): A Serial Optical Coherence Tomography Study. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 1):1518-1528. doi: 10.1016/j.jcmg.2018.08.024. Epub 2018 Dec 12. PMID 30553686
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Koskinas KC, Gencer B, Nanchen D, Branca M, Carballo D, Klingenberg R, Blum MR, Carballo S, Muller O, Matter CM, Luscher TF, Rodondi N, Heg D, Wilhelm M, Raber L, Mach F, Windecker S. Eligibility for PCSK9 inhibitors based on the 2019 ESC/EAS and 2018 ACC/AHA guidelines. Eur J Prev Cardiol. 2021 Mar 23;28(1):59-65. doi: 10.1177/2047487320940102. Epub 2020 Jul 20. PMID 33755142
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Nicholls SJ, Kataoka Y, Nissen SE, Prati F, Windecker S, Puri R, Hucko T, Aradi D, Herrman JR, Hermanides RS, Wang B, Wang H, Butters J, Di Giovanni G, Jones S, Pompili G, Psaltis PJ. Effect of Evolocumab on Coronary Plaque Phenotype and Burden in Statin-Treated Patients Following Myocardial Infarction. JACC Cardiovasc Imaging. 2022 Jul;15(7):1308-1321. doi: 10.1016/j.jcmg.2022.03.002. Epub 2022 Mar 16. PMID 35431172
- [Background] Raber L, Ueki Y, Otsuka T, Losdat S, Haner JD, Lonborg J, Fahrni G, Iglesias JF, van Geuns RJ, Ondracek AS, Radu Juul Jensen MD, Zanchin C, Stortecky S, Spirk D, Siontis GCM, Saleh L, Matter CM, Daemen J, Mach F, Heg D, Windecker S, Engstrom T, Lang IM, Koskinas KC; PACMAN-AMI collaborators. Effect of Alirocumab Added to High-Intensity Statin Therapy on Coronary Atherosclerosis in Patients With Acute Myocardial Infarction: The PACMAN-AMI Randomized Clinical Trial. JAMA. 2022 May 10;327(18):1771-1781. doi: 10.1001/jama.2022.5218. PMID 35368058
- [Background] Gao F, Wang ZJ, Ma XT, Shen H, Yang LX, Zhou YJ. Effect of alirocumab on coronary plaque in patients with coronary artery disease assessed by optical coherence tomography. Lipids Health Dis. 2021 Sep 12;20(1):106. doi: 10.1186/s12944-021-01528-3. PMID 34511134
- [Result] Liu S, Wang P, Liu C, Jin M, Wan J, Hou J, Yang Y, Wang D, Liu Z, Fu Z. Effect of PCSK9 antibodies on coronary plaque regression and stabilization derived from intravascular imaging in patients with coronary artery disease: A meta-analysis. Int J Cardiol. 2023 Dec 1;392:131330. doi: 10.1016/j.ijcard.2023.131330. Epub 2023 Sep 4. PMID 37666281